CLINICAL TRIAL: NCT02215915
Title: Intravascular Ultrasound Guided Drug Eluting Stents Implantation in "All-comers" Coronary Lesions （ULTIMATE Trial）
Acronym: ULTIMATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Shaoliang Chen, Director of Cardiology and Cath Lab, Vice President of Nanjing First Hospital, Nanjing Medical University, Nanjing First Hospital, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20140729
Record Dates: First submitted 2014-08-08; First posted 2014-08-13 (Estimated); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Coronary Artery Disease
Keywords: Percutaneous coronary intervention; Drug-eluting stent; Intravascular ultrasound
MeSH Terms: conditions — Coronary Artery Disease | interventions — Cerebral Angiography; Ultrasonography, Interventional

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IVUS guided DES implantation (Experimental): Stent size and length were selected by online IVUS measurements, and adjunct high-pressure dilation was performed according to the discretion of operators based on the IVUS criteria for stent optimization.
  Interventions: Procedure: IVUS; Procedure: DES implantation
- Angiography guided DES implantation (Active Comparator): Stent size and length were chosen by visual estimation, and adjunct high-pressure dilation was performed if an optimal result was not achieved, which was defined as angiographic residual diameter stenosis 20% and absence of angiographically detected dissection.
  Interventions: Procedure: Angiography; Procedure: DES implantation

INTERVENTIONS:
Procedure: Angiography — The size and number of stents and post-dilation will be determined on physician's discrete within the range allowed in this study protocol. All procedure will be performed according to current standard technique. Additional stent implantation or post dilation will be allowed according to attending physician's discrete. IVUS will be not used in this arm.
  Arms: Angiography guided DES implantation
Procedure: IVUS — The size and number of stents and post-dilation will be determined on physician's discrete within the range allowed in this study protocol. All procedure will be performed according to current standard technique. IVUS will be used to assess the anatomic characteristics of lesion and determine appropriate stent size and length. Additional stent implantation or post dilation will be allowed according to attending physician's discrete based on IVUS results.
  Other Names: Intravascular ultrasound
  Arms: IVUS guided DES implantation
Procedure: DES implantation
  Other Names: Percutaneous coronary drug-eluting stents implantation

SUMMARY:
A number of 1448 patients scheduled for elective percutaneous coronary intervention (PCI) with a native coronary stenosis suitable for DES implantation and IVUS imaging are openly randomized 1:1 to either IVUS guidance or angiographic guidance groups.

DETAILED DESCRIPTION:
The study is prospectively conducted at 8 high-volume PCI centers in China with IVUS expertise. Clinic follow-up are planned in all patients 12 months after implantation of drug eluting stents. Primary endpoint is target vessel failure. The study is powered for primary endpoint, which are likely to reach significance at the level P < 0.05 even at a follow-up drop-out rate up to 10%.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures;
* Men and women 18 years and older;.
* Established indication to PCI according to the guidelines of American Heart Association and American College of Cardiology;
* Native coronary lesion suitable for drug-eluting stent placement and IVUS imaging.

Exclusion Criteria:

* Pregnancy and breast feeding mother;
* Co-morbidity with an estimated life expectancy of < 50 % at 12 months;
* Scheduled major surgery in the next 12 months;
* Inability to follow the protocol and comply with follow-up requirements or any other reason that the investigator feels would place the patient at increased risk;
* Previous enrolment in this study or treatment with an investigational drug or device under another study protocol in the past 30 days;
* Known allergy against ticagrelor, or against clopidogrel, or aspirin History of major hemorrhage (intracranial, gastrointestinal, etc.);
* Chronic total occlusion lesion in either LAD, or LCX or RCA not re-canalized;
* Severe calcification needing rotational atherectomy；
* Patient with STEMI (within 24-hour from the onset of chest pain to admission).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1448 (Actual)
Dates: Start 2014-08-01 (Actual); Primary Completion 2017-05-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Target Vessel Failure | 12 months
  The occurrence of cardiac death, target vessel myocardial infraction and target vessel revascularization.

SECONDARY OUTCOMES:
Mortality | 12 months
  the occurrence of 1-year all cause death
Cardiac death | 12 months
  Death that could not be attributed to a noncardiac etiology was considered cardiac death.
Myocardial infarction | 12 months
  Myocardial infarction was diagnosed by electrocardiographic changes and/or a rise and fall of creatine kinase-myocardial band fraction in the presence of ischemic symptoms.
Target vessel revascularization | 12 months
  Target vessel revascularization was defined as repeated revascularization by PCI or surgery of the target vessel.
Target lesion revascularization | 12 months
  Target lesion revascularization was defined as any revascularization procedure performed at the site of the treated lesion associated with clinical and/or objective evidence of inducible myocardial ischemia.

OTHER OUTCOMES:
Stent thrombus | 12 months
  Stent thrombus was classified as definite, probable, or possible, according to the definitions provided by the Academic Research Consortium (ARC).Regarding timing, ST was defined as early (<30 days), late (30 days to 1 year), or too late (>1 year).

CONTACTS AND LOCATIONS:
Overall Officials: Shaoliang Chen, MD, Principal Investigator — Nanjing First Hospital, Nanjing Medical University
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee SY, Zhang JJ, Mintz GS, Hong SJ, Ahn CM, Kim JS, Kim BK, Ko YG, Choi D, Jang Y, Kan J, Pan T, Gao X, Ge Z, Chen SL, Hong MK. Procedural Characteristics of Intravascular Ultrasound-Guided Percutaneous Coronary Intervention and Their Clinical Implications. J Am Heart Assoc. 2022 Jul 19;11(14):e025258. doi: 10.1161/JAHA.122.025258. Epub 2022 Jul 15. PMID 35861828
- [Derived] Gao XF, Ge Z, Kong XQ, Kan J, Han L, Lu S, Tian NL, Lin S, Lu QH, Wang XY, Li QH, Liu ZZ, Chen Y, Qian XS, Wang J, Chai DY, Chen CH, Pan T, Ye F, Zhang JJ, Chen SL; ULTIMATE Investigators. 3-Year Outcomes of the ULTIMATE Trial Comparing Intravascular Ultrasound Versus Angiography-Guided Drug-Eluting Stent Implantation. JACC Cardiovasc Interv. 2021 Feb 8;14(3):247-257. doi: 10.1016/j.jcin.2020.10.001. Epub 2020 Oct 29. PMID 33541535
- [Derived] Zhang J, Gao X, Ge Z, Han L, Lu S, Qian X, Li Q, Lu Q, Chen C, Chen SL; ULTIMATE Investigators. Impact of intravascular ultrasound-guided drug-eluting stent implantation on patients with chronic kidney disease: Results from ULTIMATE trial. Catheter Cardiovasc Interv. 2019 Jun 1;93(7):1184-1193. doi: 10.1002/ccd.28308. Epub 2019 May 22. PMID 31116913
- [Derived] Zhang J, Gao X, Kan J, Ge Z, Han L, Lu S, Tian N, Lin S, Lu Q, Wu X, Li Q, Liu Z, Chen Y, Qian X, Wang J, Chai D, Chen C, Li X, Gogas BD, Pan T, Shan S, Ye F, Chen SL. Intravascular Ultrasound Versus Angiography-Guided Drug-Eluting Stent Implantation: The ULTIMATE Trial. J Am Coll Cardiol. 2018 Dec 18;72(24):3126-3137. doi: 10.1016/j.jacc.2018.09.013. Epub 2018 Sep 24. PMID 30261237